CLINICAL TRIAL: NCT01436487
Title: Double-Blind, Randomized, Placebo-Controlled Phase 2 Safety and Efficacy Trial of MultiStem® in Adults With Ischemic Stroke
Brief Title: Study to Examine the Effects of MultiStem in Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B01-02
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; adult stem cells
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Low dose MultiStem or Placebo
  Interventions: Biological: MultiStem; Biological: Placebo
- Cohort 2 (Experimental): High dose MultiStem or Placebo
  Interventions: Biological: MultiStem; Biological: Placebo
- Cohort 3 (Experimental): Highest, safe MultiStem dose (from Cohorts 1 and 2) or Placebo
  Interventions: Biological: MultiStem; Biological: Placebo

INTERVENTIONS:
Biological: MultiStem — single infusion 1-2 days following ischemic stroke
Biological: Placebo — single infusion 1-2 days following ischemic stroke

SUMMARY:
A study to examine the safety and potential effectiveness of the adult stem cell investigational product, MultiStem, in adults who have suffered an ischemic stroke. The hypothesis is that MultiStem will be safe and provide benefit following an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 83 years of age (inclusive)
* Clinical diagnosis of cortical cerebral ischemic stroke
* Occurrence of a moderate to moderately severe stroke

Exclusion Criteria:

* Presence of a lacunar or a brainstem infarct
* Reduced level of consciousness
* Major neurological event such as stroke or clinically significant head trauma within 6 months of study

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
frequency of dose limiting adverse events | 7 days
Stroke recovery based on global test analysis including modified Rankin Scale (mRS), NIHSS, and Barthel Index (BI) | 90 days

SECONDARY OUTCOMES:
proportion of subjects with a mRS score of less than or equal to 2 | 90 days
change in functional outcome throughout range of mRS scores | 90 days
changes in outcome measures (mRS, NIHSS, BI) over time | 365 days
proportion of subjects with an excellent functional outcome | 90 days
  * mRS score = 0 to 1; and
  * NIHSS score = 0 to 1; and
  * Barthel Index score = greater than or equal to 95
frequency of adverse events | 365 days
change in vital signs | 365 days
change in safety labs | 365 days
frequency of secondary infections | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Mays, PhD, Study Director — Healios K.K.
Locations (32):
- United States (26):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Georgia Regents University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Boston University, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - The Pennsylvania State University, Hershey, Pennsylvania
  - Hospital for the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- United Kingdom (6):
  - University of Glasgow - Western Infirmary, Glasgow
  - University of Glasgow - Southern General Hospital, Glasgow
  - St. Georges Healthcare NHS Trust, London
  - University College London Hospitals - Thames Stroke Research Network, London
  - The Newcastle upon Tyne Hospitals, NHS Foundation Trust, Newcastle upon Tyne
  - University Hospital of North Staffordshire, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess DC, Wechsler LR, Clark WM, Savitz SI, Ford GA, Chiu D, Yavagal DR, Uchino K, Liebeskind DS, Auchus AP, Sen S, Sila CA, Vest JD, Mays RW. Safety and efficacy of multipotent adult progenitor cells in acute ischaemic stroke (MASTERS): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2017 May;16(5):360-368. doi: 10.1016/S1474-4422(17)30046-7. Epub 2017 Mar 17. PMID 28320635